CLINICAL TRIAL: NCT00364260
Title: A Study to Determine the Impact of Hemoglobin Maintenance and Other Interventional Strategies to Prevent or Delay the Progression of Left Ventricular Mass Growth in Subjects With Early Renal Insufficiency.
Brief Title: A Safety and Efficacy Study for Epoetin Alfa in Pre-dialysis Subjects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR002056
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Anemia; Kidney Failure; Left Ventricular Hypertrophy
Keywords: Anemia; epoetin alfa
MeSH Terms: conditions — Anemia; Renal Insufficiency; Hypertrophy, Left Ventricular | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to determine if using Eprex, to maintain hemoglobin within the normal range, will prevent or delay the progression of left ventricular mass growth.

DETAILED DESCRIPTION:
Cardiovascular disease continues to be the major cause of morbidity and mortality in subjects with renal (kidney) disease. Left ventricular hypertrophy (LVH) has been correlated with a high risk of cardiac and all cause mortality. In the renal population , many factors have been shown to be important in the development of LVH, including anemia. This is a multicentre, open, controlled, randomized trial to determine if maintaining hemoglobin within the normal range delays the progress of left ventricular mass growth. Additionally, this study will evaluated the safety of maintaining hemoglobin within the normal range in pre-dialysis subjects. The trial duration is 24 months. Subjects randomized to the treatment arm will receive Eprex therapy to maintain hemoglobin between 120-140 g/L. Subjects randomized to the control arm will not receive any treatment unless their hemoglobin falls to less than or equal to 90 g/L. Those subjects will then be treated to maintain their hemoglobin between 90-105 g/L. The subjects were to receive injections of Eprex once weekly to maintain hemoglobin levels within the target range for the arm to which they were randomized. The subjects were to receive treatment for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients have had a decrease in hemoglobin >= 10 g/L within the past 12 months and a current hemoglobin level between 110-135 g/L (men) and 100-135 g/L (women) OR a hemoglobin level between 115-125 g/L (men) and 110-120 g/L (women)
* Have a calculated creatinine clearance <80 mL/min and >15 mL/min

Exclusion Criteria:

* No uncontrolled hypertension (diastolic blood pressure>= 105 mm Hg on average for the previous month)

No unstable angina or cardiac procedure within the past 12 months or a planned procedure

* No myocardial infarction with the past 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 1997-12; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
The change in left ventricular mass index from baseline to 24 months as measured by 2-dimensional targeted M-mode echocardiography.

SECONDARY OUTCOMES:
The difference in renal function (calculated creatinine clearance) between groups at 24 months; The functional cardiac status (NYHA/CCS classification) between groups at 24 months;The change in SF-36 scores between groups from baseline to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- [Result] Levin A, Djurdjev O, Thompson C, Barrett B, Ethier J, Carlisle E, Barre P, Magner P, Muirhead N, Tobe S, Tam P, Wadgymar JA, Kappel J, Holland D, Pichette V, Shoker A, Soltys G, Verrelli M, Singer J. Canadian randomized trial of hemoglobin maintenance to prevent or delay left ventricular mass growth in patients with CKD. Am J Kidney Dis. 2005 Nov;46(5):799-811. doi: 10.1053/j.ajkd.2005.08.007. PMID 16253719